CLINICAL TRIAL: NCT02605590
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose and Multiple Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of AIR-DNase When Administered by Inhalation to Healthy Adult Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics Study of AIR DNAse Administered by Inhalation to Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protalix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PB-110-CF01
Record Dates: First submitted 2015-11-10; First posted 2015-11-16 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Cystic Fibrosis (CF)
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1.25 mg (Experimental): Part 1: single inhaled dose of 1.25 mg AIR-DNase followed by Part 2: once daily inhaled dose of 1.25 mg AIR DNase for 5 consecutive days.
  Interventions: Drug: AIR DNase
- 2.5 mg (Experimental): Part 1: single inhaled dose of 2.5 mg AIR-DNase followed by Part 2: once daily inhaled dose of 2.5 mg AIR DNase for 5 consecutive days.
  Interventions: Drug: AIR DNase
- 5 mg (Experimental): Part 1: single inhaled dose of 5 mg AIR-DNase followed by Part 2: once daily inhaled dose of 5 mg AIR DNase for 5 consecutive days.
  Interventions: Drug: AIR DNase
- Placebo (Placebo Comparator): Placebo comparator for each of the dose levels, administered accordingly as single inhaled dose in Part 1 followed by once daily inhaled dose for 5 consecutive days in Part 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIR DNase
  Arms: 1.25 mg; 2.5 mg; 5 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will be performed to assess the safety, tolerability and PK of escalating inhaled AIR-DNase doses administered as a single dose followed by multiple doses for 5 consecutive days in healthy subjects.

A thorough review of safety data will be conducted after completion of each dose level per subject and prior to both, moving to the next dose level in Part 1 and commencement of the multiple dose Part 2.

DETAILED DESCRIPTION:
This is a Phase I study to evaluate the safety, tolerability and pharmacokinetics of inhaled AIR DNase in healthy volunteers. Up to 18 healthy males subjects (age 18 -55 inclusive) will be randomized to one of three dose cohorts (up to 6 subjects per cohort), receiving AIR DNase doses equivalent to 1.25 mg, 2.5mg or 5 mg or placebo in accordance. Subjects randomized to one of the cohorts will receive either active of placebo as single dose, in continuation, following safety assessments, will receive multiple doses, once daily for 5 consecutive days. Subjects will remain at the clinical center for 8 hours after the single administration of AIR DNase/placebo including PK sampling. During the multiple dosing subjects will arrive at the clinical center daily for AIR DNase/placebo administrations and study procedures and remain at the site for 4 hours post dosing.

Follow up visits will be performed 7±2 days following single administration and 7±2 days following the last administration of the multiple phase.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who understands the study procedures and provides written informed consent to participate in the study.
2. Healthy, male, 18-55 years of age, inclusive
3. Non smoker, by declaration, for at least 6 months prior to screening
4. Body mass index (BMI) ≥ 18.5 and ≤ 29.0 kg/m2 at screening.
5. Healthy individual with no clinically significant findings in: medical history, physical examination, laboratory profiles , vital signs, 12-lead ECG
6. Spirometry results within normal ranges.
7. A subject, whose female co-partner is of child-bearing potential, must agree to use two medically acceptable methods of contraception throughout the study.

Exclusion Criteria:

1. History of asthma, any chronic pulmonary disease, recurrent pneumonia, allergic rhinitis.
2. History of any illness or medical condition (including psychiatric) that might confound the results of the study or poses an additional risk to the subject by his participation in the study.
3. Any acute illness (e.g. acute infection) within 48 hours prior to the study drug administration, which is considered of significance by the Investigator.
4. Known contraindication, hypersensitivity and/or allergy to any drug.
5. History of adverse reactions during aerosol delivery of any medicinal product.
6. History or presence of alcoholism or drug abuse within the past 2 years prior to screening.
7. Positive urine drug of abuse test result prior to first dosing.
8. Positive breath alcohol test on admission to the CRC prior to first dosing.
9. Positive results at screening for HIV, HBsAg, or HCV Ab.
10. Sitting blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
11. Sitting heart rate is lower than 45 beats per minute (bpm) or higher than 99 bpm at screening.
12. Use of any prescription or over-the-counter medications, including vitamins, herbal, or dietary supplements within 14 days prior to dosing. Paracetamol, up to 2g /day is allowed up to 24 hours prior to dosing.
13. Donation of blood within 90 days prior to dosing.
14. Donation of bone marrow within the last 6 months prior to dosing.
15. Participation in another clinical trial within 90 days prior to dosing in which a study drug has been administered.
16. Subject is mentally or legally incapacitated or has significant emotional problems or is unable to communicate well with the investigators and CRC staff (i.e., language problem, poor mental development or impaired cerebral function).

    -

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Adverse events following inhaled single dose (SD) of AIR-DNase | 10 days
  Adverse events from subject reporting or other assessments
Adverse events following inhaled multiple doses (MD) of AIR-DNase | 14 days
  Adverse events from subject reporting or other assessments

SECONDARY OUTCOMES:
Area under the curve | 4 hours
  AIR DNase concentrations measured at 0, 0.25, 0.5, 0.75, 1, 1.5, 2, and 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Einat Almon, PhD, Study Director — Protalix Ltd.
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel